CLINICAL TRIAL: NCT06091176
Title: A Multicenter, Randomized, Parallel-Group, Single-Blind Study to Compare the Efficacy and Safety of Amicomed®, for the Management of Essential Hypertension
Brief Title: Assessment of Efficacy and Safety of Amicomed®, for the Management of Essential Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newel Health SRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NWL-AMD-CS-001
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Essential Hypertension; Primary Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Subjects assigned to ID1 treatment arm will receive Amicomed® for 90 days, together with Usual Care (UC) procedures.
  Interventions: Device: Amicomed®; Other: Usual Care
- Arm 2 (Placebo Comparator): Subjects assigned to ID2 treatment arm, will receive a digital Placebo, together with UC for 90 days.
  Interventions: Device: Digital Placebo; Other: Usual Care

INTERVENTIONS:
Device: Amicomed® — This app helps users track their blood pressure readings over time with analysis and history features. It generates graphs and charts to display trends and patterns, and users can set reminders to take blood pressure readings. Additionally, the app offers personalized recommendations for lifestyle, including personalized diet plans, and physical exercise programs based on the user's information. Using cognitive-behavioral techniques and motivational levers, the app helps users overcome barriers to lifestyle changes and provides personalized feedback and coaching. It also includes a database of evidence-based strategies for behavior change, and users can receive notifications, reminders, and rewards to stay motivated.
  Arms: Arm 1
Device: Digital Placebo — Subjects will be provided with a white label mobile app, which allows to (1) add blood pressure measurements, (2) access the history of recorded measurements. No notification system will be implemented.
  Arms: Arm 2
Other: Usual Care — Usual Care (UC): Subjects assigned to control group will receive care as usual care, including self-monitoring indications.

SUMMARY:
This is a multicenter, randomized, single-blind, parallel-group study to evaluate the efficacy and safety of Amicomed® compared with Usual Care (UC) over a 24-week treatment period in subjects with essential hypertension (mean, home based systolic blood pressure (SBP) ≥ 140 and/or diastolic blood pressure DBP ≥ 90 mm Hg on Day 1).

DETAILED DESCRIPTION:
Amicomed is a Digital therapeutics service and program for BP management and reduction. The key features of Amicomed include:

1. an automatic, expert system based, finite-machine AI algorithm for assessing the evolution of blood pressure levels,
2. an automatic, expert system based, finite-machine AI algorithm for generating and delivering a detailed lifestyle program (dietary and physical activity) starting from the general lifestyle suggestions of the hypertension and cardiovascular prevention guidelines and producing a truly personalized program.
3. a behavioral strategy embedded into the app to increase adherence and persistence into the program.

The Amicomed Digital Therapeutics Service and App for hypertension management and intervention has been shown to significantly improve BP levels in case-control studies .These initial results demonstrated a 5mmHg systolic BP reduction across all Amicomed subscribers and 7.9 mmHg systolic BP reduction in subject with >= stage 1 hypertension. Comparable reduction of diastolic BP was also achieved.

The aim of this study is to investigate the long-term efficacy of the Amicomed® Digital Therapeutics Program, compared to Usual Care, in reducing Systolic and Diastolic Blood Pressure in subjects with primary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with age ≥ 18 years
* Diagnosed with essential hypertension and exhibiting a mean home-based SBP ≥ 140 and/or DBP > 90mm Hg, i.e., Grade I Hypertension .
* Disease duration: 12 (+/-) 3 months
* Unmedicated, or currently treated by a stable regimen for hypertension with sub-optimal response to usual care treatments (Delta SBP < 5 mm Hg; and/or Delta DBP < 5 mm Hg)
* Not participating in physical exercise or dietary programs during the last 12 months from Visit 1.
* Willing and able to return for all clinic visits and to complete all study-required procedures
* Able to use the app, [self-report compliance over 80%]. Compliance is defined as the capacity to provide at least 6 BP measurements per week during the beginning, middle and end week of the 24 weeks program.

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the study period
* Use of medications that may interfere with the study intervention
* Severe kidney or liver disease
* Active cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Home Blood Pressure Monitoring - Systolic Blood Pressure | Baseline to Week 12
  The primary endpoint is change from baseline to Week 12 in trough (approximately 7 days before the previous visit) Home BP SBP.
  Home BP is the average of all BP readings performed with a semiautomatic, validated BP monitor, for at least 3 days and preferably for 6-7 consecutive days before each clinic visit, with readings in the morning and the evening, taken in a quiet room after 5 min of rest, with the patient seated with their back and arm supported. Two measurements should be taken at each measurement session, performed 1-2 min apart.
  The primary endpoints will be collected using dedicated BP monitoring devices. Measurements taken for the purpose of efficacy assessment will not be reported to, nor shared or collected through the Investigational Device ID1.
Change in Home Blood Pressure Monitoring - Dyastolic Blood Pressure | Baseline to Week 12
  The primary endpoint is change from baseline to Week 12 in trough (approximately 7 days before the previous visit) Home BP SBP.
  Home BP is the average of all BP readings performed with a semiautomatic, validated BP monitor, for at least 3 days and preferably for 6-7 consecutive days before each clinic visit, with readings in the morning and the evening, taken in a quiet room after 5 min of rest, with the patient seated with their back and arm supported. Two measurements should be taken at each measurement session, performed 1-2 min apart.
  The primary endpoints will be collected using dedicated BP monitoring devices. Measurements taken for the purpose of efficacy assessment will not be reported to, nor shared or collected through the Investigational Device ID1.

SECONDARY OUTCOMES:
The change from baseline to Week 24 in trough Home BP Systolic Blood Pressure | Baseline to Week 24
  Change from baseline to Week 24 in trough (approximately 7 days before the previous visit) Home BP SBP.
  Home BP is the average of all BP readings performed with a semiautomatic, validated BP monitor, for at least 3 days and preferably for 6-7 consecutive days before each clinic visit, with readings in the morning and the evening, taken in a quiet room after 5 min of rest, with the patient seated with their back and arm supported. Two measurements should be taken at each measurement session, performed 1-2 min apart.
  The endpoints will be collected using dedicated BP monitoring devices. Measurements taken for the purpose of efficacy assessment will not be reported to, nor shared or collected through the Investigational Device ID1.
The change from baseline to Week 24 in trough Home BP Diastolic Blood Pressure | Baseline to Week 24
  Change from baseline to Week 24 in trough (approximately 7 days before the previous visit) Home BP DBP.
  Home BP is the average of all BP readings performed with a semiautomatic, validated BP monitor, for at least 3 days and preferably for 6-7 consecutive days before each clinic visit, with readings in the morning and the evening, taken in a quiet room after 5 min of rest, with the patient seated with their back and arm supported. Two measurements should be taken at each measurement session, performed 1-2 min apart.
  The endpoints will be collected using dedicated BP monitoring devices. Measurements taken for the purpose of efficacy assessment will not be reported to, nor shared or collected through the Investigational Device ID1.
Percentage of responders at Week 12 Home BP SBP <140 mm Hg and/or reduction of ≥5 mm Hg from baseline. | Baseline to Week 12
  Percentage of responders who show at Week 12 Home BP SBP <140 mm Hg and/or a reduction of ≥5 mm Hg from baseline.
Percentage of responders at Week 24 Home BP SBP <140 mm Hg and/or reduction of ≥5 mm Hg from baseline. | Baseline to Week 24
  Percentage of responders who show at Week 24 Home BP SBP <140 mm Hg and/or a reduction of ≥5 mm Hg from baseline.
Percentage of responders at Week 12 Home BP DBP <90 mm Hg and/or reduction of ≥5 mm Hg from baseline. | Baseline to Week 12
  Percentage of responders who show at Week 12 Home BP DBP <90 mm Hg and/or a reduction of ≥5 mm Hg from baseline.
Percentage of responders at Week 24 Home BP DBP <90 mm Hg and/or reduction of ≥5 mm Hg from baseline. | Baseline to Week 24
  Percentage of responders who show at Week 24 Home BP DBP <90 mm Hg and/or reduction of ≥5 mm Hg from baseline.
Percentage of subjects achieving target blood pressure Home BP SBP <140 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP SBP <140 mm Hg.
Percentage of subjects achieving target blood pressure Home BP DBP <90 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP SBP <140 mm Hg.
Percentage of subjects achieving target blood pressure Home BP SBP <140 mm Hg and DBP <90 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP SBP <140 mm Hg and DBP <90 mm Hg.
Percentage of subjects achieving target blood pressure Home BP DBP <80 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP DBP <80 mm Hg.
Percentage of subjects achieving target blood pressure Home BP SBP <130 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP SBP <130 mm Hg.
Percentage of subjects achieving target blood pressure Home BP SBP <130 mm Hg and DBP <80 mm Hg. | Baseline to Week 12
  Percentage of subjects achieving target blood pressure Home BP SBP <130 mm Hg and DBP <80 mm Hg.
Mean changes in weight | Baseline to Week 12; Baseline to Week 24
  Mean changes in weight, expressed in Kilograms (Kg)
Mean changes in BMI | Baseline to Week 12; Baseline to Week 24
  Mean changes in Body Mass Index
Mean changes in waist circumference | Baseline to Week 12; Baseline to Week 24
  Mean changes in waist circumference, expressed in centimeters (cm).
Mean change in points obtained by salt intake check sheet. | Baseline to Week 12; Baseline to Week 24
  Mean change in points obtained by salt intake check sheet.
Amicomed(R) app usage rate | Baseline to Week 12; Baseline to Week 24
  Amicomed(R) app usage rate: Percentage of usage of Amicomed(R) app
Amicomed(R) progress of app educational programs | Baseline to Week 12; Baseline to Week 24
  Amicomed(R) progress of app educational programs
Rate of home BP measurements | Baseline to Week 12; Baseline to Week 24
  Weekly Rate of home BP measurements
Malfunctions of the investigational medical device | Baseline to Week 12; Baseline to Week 24
  Frequency of reported malfunctions of the investigational medical device
Percentage of subjects on medication for Hypertension | Baseline to Week 12; Baseline to Week 24
  Percentage of subjects on medication for Hypertension

OTHER OUTCOMES:
Any adverse events including device-related adverse events. | Baseline to Week 12; Baseline to Week 24
  Any adverse events including device-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Cianflone, MD, PhD, Study Chair — Newel Health SRL

IPD SHARING:
Plan to Share IPD: No